CLINICAL TRIAL: NCT00210522
Title: A Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy, Safety, and Tolerability of RWJ-333369 as Adjunctive Therapy in Subjects With Refractory Partial Seizures (Protocol 333369-EPY-2003 [Double-blind] and Protocol 333369-EPY-2006 [Open-label Extension])
Brief Title: An Open-Label Extension Study of the Effectiveness and Safety of the Investigational Compound RWJ-333369 in Patients With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002191
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Epilepsy; Epilepsies, Partial
Keywords: RWJ-333369; Anticonvulsants; Epilepsy; Refractory partial epilepsy; Seizure disorder; Antiepileptic drugs
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

ARMS (1):
- 001 (Experimental): RWJ 333369 Open-Label Extension: One 200 mg to 600mg tablet taken twice daily (up to a maximum of 1200mg/day) up to 1 year or the time that RWJ-333369 is available by prescription or the study is terminated by Sponsor.
  Interventions: Drug: RWJ 333369

INTERVENTIONS:
Drug: RWJ 333369 — Open-Label Extension: One 200 mg to 600mg tablet taken twice daily (up to a maximum of 1200mg/day) up to 1 year or the time that RWJ-333369 is available by prescription or the study is terminated by Sponsor.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the novel compound RWJ-333369 in reducing the frequency of seizures in patients with epilepsy.

DETAILED DESCRIPTION:
333369EPY2006 is the open-label extension study that follows the double-blind study 333369EPY2003. In an open label study such as 333369EPY2006, both the physician and the patient know the name of the assigned study medication. In a double blind study such as 333369EPY2003, neither the physician nor the patient knows the name of the assigned study medication. Patients who complete the double-blind treatment phase of study 333369EPY2003 will be eligible to enter the open-label extension study during which patients will transition through a blinded period to an open-label period with carisbamate (also referred to as RWJ-333369). RWJ-333369 is a new chemical compound with anticonvulsant activity that is currently under investigation as a treatment for epilepsy. Patients electing to enter the open-label extension phase will be supplied with both open-label carisbamate (RWJ-333369) and blinded study medication for the transition phase. During this transition phase (approximately 3 weeks in length), the patient's dose of double-blind study drug will be gradually reduced and stopped and treatment with open-label RWJ-333369 will be started. Throughout the remainder of the open label extension phase, investigators will be allowed to make further adjustments of the dosage and schedule of carisbamate, including independent adjustment of the morning and evening doses, but a dosage of 1,200 mg/day may not be exceeded and increases in dosage must be in increments of no more than 200 mg/day. After 12 months of participation in the open-label extension study, patients who, in the judgment of the investigator, continue to benefit from treatment with RWJ-333369 may continue to receive the drug with follow up clinic visits every 3 months until RWJ 333369 is available by prescription or the program is terminated by the sponsor. RWJ-333369 (100, 300, 800, or 1,600 milligrams per day) administered orally in 2 equally divided doses for up to 16 weeks of double-blind treatment followed by the option to continue RWJ-333369 treatment in an open-label study for at least 1 year, then until drug is available or production ceases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must complete Visit 8 (Day 112) of the double-blind treatment phase of Study EPY-2003 to be eligible for entry into the open-label treatment phase of Study EPY-2006.

Exclusion Criteria:

* Patients who have seizures that cannot be quantitated accurately
* Patients with a history of nonepileptic seizures, serious systemic disease, progressive neurologic disorder, a major psychiatric disorder, status epilepticus in the past 3 months, vagal nerve stimulation discontinuation within the past 3 months
* Patients with a history of drug or alcohol abuse within the past 2 years
* Patients currently taking felbamate, vigabatrin, or tricyclic antidepressants
* and patients who are pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2005-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 1 year or until carisbamate is available by prescription or the study is terminated by the sponsor
Clinical laboratory test values | Up to 1 year or until carisbamate is available by prescription or the study is terminated by the sponsor
12-lead ECG recordings | Up to 1 year or until carisbamate is available by prescription or the study is terminated by the sponsor
Vital sign measurements | Up to 1 year or until carisbamate is available by prescription or the study is terminated by the sponsor

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Faught E, Holmes GL, Rosenfeld WE, Novak G, Neto W, Greenspan A, Schmitt J, Yuen E, Reines S, Haas M. Randomized, controlled, dose-ranging trial of carisbamate for partial-onset seizures. Neurology. 2008 Nov 11;71(20):1586-93. doi: 10.1212/01.wnl.0000334751.89859.7f. PMID 19001248